CLINICAL TRIAL: NCT06900907
Title: Comparison of the Effects of Ozone Therapy, Hyaluronic Acid, Methylprednisolone, and Low-Level Laser Therapy on Pain, Edema, and Trismus Following Surgical Extraction of Impacted Lower Third Molars
Brief Title: Comparison of the Effects of Protocols Applied After Surgical Extraction of Impacted Mandibular Third Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batman University (Other)
Responsible Party: Principal Investigator, Rojdan Ferman GÜNEŞ UYSAL, Assistant professor, Batman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BatmanU-DF-RFGU-03; DİŞ.15.023 (Other Grant/Funding Number: Dicle University Scientific Research Projects Coordination)
Record Dates: First submitted 2025-03-22; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Tooth Impaction | {Tooth} | Dental; Corticosteroid; Hyaluronic Acid; Ozone; Laser Therapy
MeSH Terms: conditions — Tooth, Impacted | interventions — Lasers, Semiconductor; Hyaluronic Acid; Ozone; Methylprednisolone; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 Laser (Experimental): In Group 1, after the extraction of the impacted third molar, a diode laser (Epic X, Biolase, USA) with a wavelength of 940 nm and power of 0.2 W was applied in non-contact mode for 25 seconds at an energy density of 10 J/cm² to the occlusal, buccal, and lingual surfaces of the extraction site.
  Interventions: Device: Diode laser
- Group 2 Hyaluronic acid (Experimental): In Group 2, after the extraction of the impacted third molar, 1 cc of high-molecular-weight hyaluronic acid gel (240 mg/100 g) (Bioplax, London, UK) was placed into the extraction socket.
  Interventions: Combination Product: Hyaluronic acid
- Group 3 Ozone (Experimental): In Group 3, after the extraction of the impacted third molar, topical ozone therapy (W&H Prozone Ozone Generator) was applied to the extraction socket for 15 seconds.
  Interventions: Combination Product: Ozone
- Group 4 Methylprednisolone (Experimental): In Group 4, in addition to the standard prescribed medication, patients received 4 mg oral methylprednisolone (Koçak Farma İlaç ve Kimya Sanayi A.Ş., Istanbul) starting immediately after surgery. It was administered three times on the first day, twice on the second day, and once on the third day.
  Interventions: Drug: Methylprednisolone
- Group 5 Control (Active Comparator): In Group 5 (control group), only the standard prescribed medication was provided.
  Interventions: Procedure: Control

INTERVENTIONS:
Device: Diode laser — A single session was applied to three points of the tooth extraction site.
  Other Names: Epic X, Biolase, USA
  Arms: Group 1 Laser
Combination Product: Hyaluronic acid — 1 cc of hyaluronic acid gel was placed into the extraction socket, followed by suturing.
  Other Names: Aftamed ®
  Arms: Group 2 Hyaluronic acid
Combination Product: Ozone — Topical ozone was applied to the extraction socket, followed by suturing.
  Other Names: W&H Prozone Ozone Generator
  Arms: Group 3 Ozone
Drug: Methylprednisolone — In addition to the standard prescribed medication, 4 mg of oral methylprednisolone was prescribed postoperatively.
  Other Names: Precort 4 mg Tablet
  Arms: Group 4 Methylprednisolone
Procedure: Control — Only the standard prescribed medication was provided.
  Arms: Group 5 Control

SUMMARY:
Following the surgical extraction of the most commonly impacted mandibular third molars, the first group was planned to receive methylprednisolone, the second group hyaluronic acid, the third group ozone therapy, the fourth group laser application, and the fifth group only the routine treatment protocol. The study comparatively evaluated the effectiveness of these five groups in preventing complications such as pain, edema, and trismus that may develop after impacted third molar surgery.

DETAILED DESCRIPTION:
The mandibular third molars are the most commonly impacted teeth in the jaws, and their surgical extraction is a frequently performed procedure in oral and maxillofacial surgery clinics. Postoperative pain, trismus, and edema, particularly within the first 48 hours after surgery, significantly impair patients' quality of life. In addition to routinely prescribed medications, various postoperative treatment methods have been explored to minimize or control these complications. Some of the methods reported in the literature include corticosteroid administration, low-level laser therapy, hyaluronic acid application at the extraction site, and ozone therapy.

Corticosteroids exert their anti-inflammatory effects by inhibiting both the function and production of certain inflammatory cells. Therefore, they have been widely used for many years to reduce complications following impacted third molar surgery. Low-level laser therapy (LLLT) has anti-inflammatory and analgesic properties, as well as a biostimulatory effect that promotes wound healing. Ozone therapy, due to its antibacterial and anti-inflammatory properties, as well as its ability to accelerate epithelial healing, has been recognized in the literature as a modern, drug-free alternative for managing postoperative complications.

Hyaluronic acid (HA) is a member of the glycosaminoglycan family found in various body tissues. Due to its numerous advantages, including the promotion of wound healing, anti-inflammatory, bacteriostatic, and osteoinductive effects, it plays a crucial role in tissue healing and the prevention of postoperative sequelae.

This study comparatively evaluates the efficacy of low-level laser therapy, hyaluronic acid, ozone therapy, and methylprednisolone in preventing complications such as pain, edema, and trismus following impacted mandibular third molar surgery, with the aim of improving patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients classified as American Society of Anesthesiologists (ASA) Class I or II
* Age range of 18-35 years
* Individuals of both genders
* Horizontally impacted teeth with the same angulation according to Winter's classification

Exclusion Criteria:

* Patients with any pathological condition around the impacted tooth
* Pregnant or breastfeeding women
* Smokers
* Individuals with allergic reactions to the adjuvants or prescribed medications used in the study
* Surgical extraction procedures exceeding 30 minutes

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
Trismus | All patient data were collected on the 3rd and 7th postoperative days by a researcher blinded to the study groups.
  Preoperative maximum mouth opening for trismus (measured as the distance between the upper right and lower right central incisors) was recorded using a Vernier caliper (Mayerbach M003, Germany)

SECONDARY OUTCOMES:
Edema | All patient data were collected on the 3rd and 7th postoperative days by a researcher blinded to the study groups.
  For edema assessment, a widely used method in the literature was applied, measuring the linear distances between the lateral canthus-gonion, tragus-pogonion, and tragus-labial commissure points using a flexible measuring tape in direct contact with the skin

OTHER OUTCOMES:
Pain Level | All patient data were collected on the 3rd and 7th postoperative days by a researcher blinded to the study groups.
  Pain levels were assessed using a visual analog scale (VAS) form, numbered from 1 to 10. For each follow-up period, patients were instructed to mark a value where 0 indicated no pain, 10 represented unbearable pain, and intermediate values reflected varying pain intensities.

CONTACTS AND LOCATIONS:
Overall Officials: Nedim GÜNEŞ, Ass.Prof., Study Chair — Dicle University
Locations (1):
- Dicle University, Diyarbakır, Sur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No